CLINICAL TRIAL: NCT04071847
Title: Abbott DBS Post-Market Study of Outcomes for Indications Over Time
Acronym: ADROIT
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10300
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Movement Disorders; Parkinson Disease; Essential Tremor; Tremor; Dystonia; Primary Dystonia; Secondary Dystonia
MeSH Terms: conditions — Movement Disorders; Parkinson Disease; Essential Tremor; Tremor; Dystonia; Dystonic Disorders | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Deep brain stimulation: Subjects implanted with an Abbott DBS system
  Interventions: Device: Deep Brain Stimulation (DBS)

INTERVENTIONS:
Device: Deep Brain Stimulation (DBS) — Deep brain stimulation therapy involves the delivery of electrical signals to targeted structures in the brain to modulate neural circuit activity, and has been used successfully for the treatment of various types of movement disorders, including Parkinson's disease (PD), disabling or essential tremor, and dystonia

SUMMARY:
The purpose of this international study is to evaluate long-term safety and effectiveness of Abbott deep brain stimulation (DBS) systems for all indications, including Parkinson's disease, essential tremor or other disabling tremor and dystonia.

DETAILED DESCRIPTION:
ADROIT is an international, prospective, multicenter, observational, post-market study intended to collect worldwide long-term safety and effectiveness data on subjects implanted with market-released Abbott DBS systems in routine clinical practice.

Subjects will be followed for 5 years after the initial programming visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is scheduled for a new implant or IPG device replacement surgery with a market-released Abbott DBS system within 180 days.
2. Subject, or a legally acceptable representative, must provide written informed consent prior to any study-related procedure.

Exclusion Criteria:

1. Subject is currently enrolled or plans to enroll in an investigational study that may confound the results of this study.
2. Subject has anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the study or to comply with follow-up requirements, or impact the scientific soundness of the study results.
3. Study center is located in the United States, and indication for DBS implant is not Parkinson's disease or disabling tremor.
4. Study center is located in the United States, and the intended lead implant location is not at, or in close proximity to, the STN, GPi, or VIM thalamus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll male and female subjects diagnosed with Parkinson's disease, essential tremor or other disabling tremor, or dystonia who are scheduled for a new implant or IPG device replacement surgery with a market-released Abbott DBS system.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-11-26 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 6 months in disease-specific motor rating scale. For subjects with Parkinson's disease, MDS-UPDRS Part III. | Baseline to 6 months
  The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) assess the severity of Parkinson's disease. This questionnaire is composed of four sections: Part I: non-motor experiences of daily living consisting of 13 questions (Part Ia is assessed by the investigator while part Ib is assessed by the subject, with or without the help of the caregiver); Part II: motor experiences of daily living consisting of 13 questions, designed to be self-administered; Part III: motor examinations consisting of 33 scores based on 18 questions with several right, left or other body distribution scores; Part IV: motor complications: consisting of 6 questions. Each item is scored from 0 to 4, where 0 indicates normal, 1 indicates slight symptoms, 2 indicates mild symptoms, 3 indicates moderate symptoms, and 4 indicates severe symptoms. The total score for each part is obtained from the sum of the corresponding item scores. Higher scores indicate greater impact of PD symptoms.
Change from baseline to1 year in disease-specific motor rating scale. For subjects with Parkinson's disease, MDS-UPDRS Part III. | Baseline to1 year
  The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) assess the severity of Parkinson's disease. This questionnaire is composed of four sections: Part I: non-motor experiences of daily living consisting of 13 questions (Part Ia is assessed by the investigator while part Ib is assessed by the subject, with or without the help of the caregiver); Part II: motor experiences of daily living consisting of 13 questions, designed to be self-administered; Part III: motor examinations consisting of 33 scores based on 18 questions with several right, left or other body distribution scores; Part IV: motor complications: consisting of 6 questions. Each item is scored from 0 to 4, where 0 indicates normal, 1 indicates slight symptoms, 2 indicates mild symptoms, 3 indicates moderate symptoms, and 4 indicates severe symptoms. The total score for each part is obtained from the sum of the corresponding item scores. Higher scores indicate greater impact of PD symptoms.
Change from baseline to 2 years in disease-specific motor rating scale. For subjects with Parkinson's disease, MDS-UPDRS Part III. | Baseline to 2 years
  The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) assess the severity of Parkinson's disease. This questionnaire is composed of four sections: Part I: non-motor experiences of daily living consisting of 13 questions (Part Ia is assessed by the investigator while part Ib is assessed by the subject, with or without the help of the caregiver); Part II: motor experiences of daily living consisting of 13 questions, designed to be self-administered; Part III: motor examinations consisting of 33 scores based on 18 questions with several right, left or other body distribution scores; Part IV: motor complications: consisting of 6 questions. Each item is scored from 0 to 4, where 0 indicates normal, 1 indicates slight symptoms, 2 indicates mild symptoms, 3 indicates moderate symptoms, and 4 indicates severe symptoms. The total score for each part is obtained from the sum of the corresponding item scores. Higher scores indicate greater impact of PD symptoms.
Change from baseline to 3 years in disease-specific motor rating scale. For subjects with Parkinson's disease, MDS-UPDRS Part III. | Baseline to 3 years
  The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) assess the severity of Parkinson's disease. This questionnaire is composed of four sections: Part I: non-motor experiences of daily living consisting of 13 questions (Part Ia is assessed by the investigator while part Ib is assessed by the subject, with or without the help of the caregiver); Part II: motor experiences of daily living consisting of 13 questions, designed to be self-administered; Part III: motor examinations consisting of 33 scores based on 18 questions with several right, left or other body distribution scores; Part IV: motor complications: consisting of 6 questions. Each item is scored from 0 to 4, where 0 indicates normal, 1 indicates slight symptoms, 2 indicates mild symptoms, 3 indicates moderate symptoms, and 4 indicates severe symptoms. The total score for each part is obtained from the sum of the corresponding item scores. Higher scores indicate greater impact of PD symptoms.
Change from baseline to 4 years in disease-specific motor rating scale. For subjects with Parkinson's disease, MDS-UPDRS Part III. | Baseline to 4 years
  The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) assess the severity of Parkinson's disease. This questionnaire is composed of four sections: Part I: non-motor experiences of daily living consisting of 13 questions (Part Ia is assessed by the investigator while part Ib is assessed by the subject, with or without the help of the caregiver); Part II: motor experiences of daily living consisting of 13 questions, designed to be self-administered; Part III: motor examinations consisting of 33 scores based on 18 questions with several right, left or other body distribution scores; Part IV: motor complications: consisting of 6 questions. Each item is scored from 0 to 4, where 0 indicates normal, 1 indicates slight symptoms, 2 indicates mild symptoms, 3 indicates moderate symptoms, and 4 indicates severe symptoms. The total score for each part is obtained from the sum of the corresponding item scores. Higher scores indicate greater impact of PD symptoms.
Change from baseline to 5 years in disease-specific motor rating scale. For subjects with Parkinson's disease, MDS-UPDRS Part III. | Baseline to 5 years
  The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) assess the severity of Parkinson's disease. This questionnaire is composed of four sections: Part I: non-motor experiences of daily living consisting of 13 questions (Part Ia is assessed by the investigator while part Ib is assessed by the subject, with or without the help of the caregiver); Part II: motor experiences of daily living consisting of 13 questions, designed to be self-administered; Part III: motor examinations consisting of 33 scores based on 18 questions with several right, left or other body distribution scores; Part IV: motor complications: consisting of 6 questions. Each item is scored from 0 to 4, where 0 indicates normal, 1 indicates slight symptoms, 2 indicates mild symptoms, 3 indicates moderate symptoms, and 4 indicates severe symptoms. The total score for each part is obtained from the sum of the corresponding item scores. Higher scores indicate greater impact of PD symptoms.
Change from baseline to 6 months in disease-specific motor rating scale. For subjects with disabling tremor, FTM-TRS. | Baseline to 6 months
  The Fahn-Tolosa-Marin Tremor Rating Scale (FTMTRS) assesses tremor severity and and consists of three parts. Part A (with a maximum score of 80) rates tremor at rest, during posture, and intentional movements for nine parts of the body, including the head, trunk and limbs; Part B (with a maximum score of 36) rates action tremor of the upper limbs, particularly while writing and pouring liquids; part C the patient rates the impact of tremor on his or her functional disability (speaking, feeding, drinking, hygiene, dressing, writing, and working) with a maximum score of 28. The total score obtained by adding the three parts of the FTM-TRS is 144, with a higher score indicating higher disease severity/disability.
  The FTM-TRS also includes one separate item dealing with global assessment of tremor-related disability, rated by both patient and examiner on a 5-point scale.
Change from baseline to 1 year in disease-specific motor rating scale. For subjects with disabling tremor, FTM-TRS. | Baseline to 1 year
  The Fahn-Tolosa-Marin Tremor Rating Scale (FTMTRS) assesses tremor severity and and consists of three parts. Part A (with a maximum score of 80) rates tremor at rest, during posture, and intentional movements for nine parts of the body, including the head, trunk and limbs; Part B (with a maximum score of 36) rates action tremor of the upper limbs, particularly while writing and pouring liquids; part C the patient rates the impact of tremor on his or her functional disability (speaking, feeding, drinking, hygiene, dressing, writing, and working) with a maximum score of 28. The total score obtained by adding the three parts of the FTM-TRS is 144, with a higher score indicating higher disease severity/disability.The FTM-TRS also includes one separate item dealing with global assessment of tremor-related disability, rated by both patient and examiner on a 5-point scale.
Change from baseline to 2 years in disease-specific motor rating scale. For subjects with disabling tremor, FTM-TRS. | Baseline to 2 years
  The Fahn-Tolosa-Marin Tremor Rating Scale (FTMTRS) assesses tremor severity and and consists of three parts. Part A (with a maximum score of 80) rates tremor at rest, during posture, and intentional movements for nine parts of the body, including the head, trunk and limbs; Part B (with a maximum score of 36) rates action tremor of the upper limbs, particularly while writing and pouring liquids; part C the patient rates the impact of tremor on his or her functional disability (speaking, feeding, drinking, hygiene, dressing, writing, and working) with a maximum score of 28. The total score obtained by adding the three parts of the FTM-TRS is 144, with a higher score indicating higher disease severity/disability.The FTM-TRS also includes one separate item dealing with global assessment of tremor-related disability, rated by both patient and examiner on a 5-point scale.
Change from baseline to 3 years in disease-specific motor rating scale. For subjects with disabling tremor, FTM-TRS. | Baseline to 3 years
  The Fahn-Tolosa-Marin Tremor Rating Scale (FTMTRS) assesses tremor severity and and consists of three parts. Part A (with a maximum score of 80) rates tremor at rest, during posture, and intentional movements for nine parts of the body, including the head, trunk and limbs; Part B (with a maximum score of 36) rates action tremor of the upper limbs, particularly while writing and pouring liquids; part C the patient rates the impact of tremor on his or her functional disability (speaking, feeding, drinking, hygiene, dressing, writing, and working) with a maximum score of 28. The total score obtained by adding the three parts of the FTM-TRS is 144, with a higher score indicating higher disease severity/disability.The FTM-TRS also includes one separate item dealing with global assessment of tremor-related disability, rated by both patient and examiner on a 5-point scale.
Change from baseline to 4 years in disease-specific motor rating scale. For subjects with disabling tremor, FTM-TRS. | Baseline to 4 years
  The Fahn-Tolosa-Marin Tremor Rating Scale (FTMTRS) assesses tremor severity and and consists of three parts. Part A (with a maximum score of 80) rates tremor at rest, during posture, and intentional movements for nine parts of the body, including the head, trunk and limbs; Part B (with a maximum score of 36) rates action tremor of the upper limbs, particularly while writing and pouring liquids; part C the patient rates the impact of tremor on his or her functional disability (speaking, feeding, drinking, hygiene, dressing, writing, and working) with a maximum score of 28. The total score obtained by adding the three parts of the FTM-TRS is 144, with a higher score indicating higher disease severity/disability. The FTM-TRS also includes one separate item dealing with global assessment of tremor-related disability, rated by both patient and examiner on a 5-point scale.
Change from baseline to 5 years in disease-specific motor rating scale. For subjects with disabling tremor, FTM-TRS. | Baseline to 5 years
  The Fahn-Tolosa-Marin Tremor Rating Scale (FTMTRS) assesses tremor severity and and consists of three parts. Part A (with a maximum score of 80) rates tremor at rest, during posture, and intentional movements for nine parts of the body, including the head, trunk and limbs; Part B (with a maximum score of 36) rates action tremor of the upper limbs, particularly while writing and pouring liquids; part C the patient rates the impact of tremor on his or her functional disability (speaking, feeding, drinking, hygiene, dressing, writing, and working) with a maximum score of 28. The total score obtained by adding the three parts of the FTM-TRS is 144, with a higher score indicating higher disease severity/disability.The FTM-TRS also includes one separate item dealing with global assessment of tremor-related disability, rated by both patient and examiner on a 5-point scale.
Change from baseline to 6 months in disease-specific motor rating scale. For subjects with dystonia (except for cervical dystonia), BFMDRS movement scale. | Baseline to 6 months
  The BFMDRS consists consists of a movement subscale and a disability subscale. The movement scale measures dystonia in nine body regions (including the eyes, mouth, speech and swallowing, neck, trunk, arms, and legs). Each domain is scored on degree of provoking factor (0=no dystonia at rest or with action to 4=dystonia present at rest) and severity factor (0=no dystonia to 4=extreme/severe dystonia). Scores are weighted yielding a total score ranging from 0 to 120. The disability scale is a functional marker consisting of parental- or self-reported daily activities (involving speech, handwriting, feeding, eating, swallowing, hygiene, dressing, and walking), with scores ranging from 0 (completely independent) to 30 (completely dependent). A higher score indicates higher disease severity/disability.
Change from baseline to 1 year in disease-specific motor rating scale. For subjects with dystonia (except for cervical dystonia), BFMDRS movement scale. | Baseline to 1 year
  The BFMDRS consists consists of a movement subscale and a disability subscale. The movement scale measures dystonia in nine body regions (including the eyes, mouth, speech and swallowing, neck, trunk, arms, and legs). Each domain is scored on degree of provoking factor (0=no dystonia at rest or with action to 4=dystonia present at rest) and severity factor (0=no dystonia to 4=extreme/severe dystonia). Scores are weighted yielding a total score ranging from 0 to 120. The disability scale is a functional marker consisting of parental- or self-reported daily activities (involving speech, handwriting, feeding, eating, swallowing, hygiene, dressing, and walking), with scores ranging from 0 (completely independent) to 30 (completely dependent). A higher score indicates higher disease severity/disability.
Change from baseline to 2 years in disease-specific motor rating scale. For subjects with dystonia (except for cervical dystonia), BFMDRS movement scale. | Baseline to 2 years
  The BFMDRS consists consists of a movement subscale and a disability subscale. The movement scale measures dystonia in nine body regions (including the eyes, mouth, speech and swallowing, neck, trunk, arms, and legs). Each domain is scored on degree of provoking factor (0=no dystonia at rest or with action to 4=dystonia present at rest) and severity factor (0=no dystonia to 4=extreme/severe dystonia). Scores are weighted yielding a total score ranging from 0 to 120. The disability scale is a functional marker consisting of parental- or self-reported daily activities (involving speech, handwriting, feeding, eating, swallowing, hygiene, dressing, and walking), with scores ranging from 0 (completely independent) to 30 (completely dependent). A higher score indicates higher disease severity/disability.
Change from baseline to 3 years in disease-specific motor rating scale. For subjects with dystonia (except for cervical dystonia), BFMDRS movement scale. | Baseline to 3 years
  The BFMDRS consists consists of a movement subscale and a disability subscale. The movement scale measures dystonia in nine body regions (including the eyes, mouth, speech and swallowing, neck, trunk, arms, and legs). Each domain is scored on degree of provoking factor (0=no dystonia at rest or with action to 4=dystonia present at rest) and severity factor (0=no dystonia to 4=extreme/severe dystonia). Scores are weighted yielding a total score ranging from 0 to 120. The disability scale is a functional marker consisting of parental- or self-reported daily activities (involving speech, handwriting, feeding, eating, swallowing, hygiene, dressing, and walking), with scores ranging from 0 (completely independent) to 30 (completely dependent). A higher score indicates higher disease severity/disability.
Change from baseline to 4 years in disease-specific motor rating scale. For subjects with dystonia (except for cervical dystonia), BFMDRS movement scale. | Baseline to 4 years
  The BFMDRS consists consists of a movement subscale and a disability subscale. The movement scale measures dystonia in nine body regions (including the eyes, mouth, speech and swallowing, neck, trunk, arms, and legs). Each domain is scored on degree of provoking factor (0=no dystonia at rest or with action to 4=dystonia present at rest) and severity factor (0=no dystonia to 4=extreme/severe dystonia). Scores are weighted yielding a total score ranging from 0 to 120. The disability scale is a functional marker consisting of parental- or self-reported daily activities (involving speech, handwriting, feeding, eating, swallowing, hygiene, dressing, and walking), with scores ranging from 0 (completely independent) to 30 (completely dependent). A higher score indicates higher disease severity/disability.
Change from baseline to 5 years in disease-specific motor rating scale. For subjects with dystonia (except for cervical dystonia), BFMDRS movement scale. | Baseline to 5 years
  The BFMDRS consists consists of a movement subscale and a disability subscale. The movement scale measures dystonia in nine body regions (including the eyes, mouth, speech and swallowing, neck, trunk, arms, and legs). Each domain is scored on degree of provoking factor (0=no dystonia at rest or with action to 4=dystonia present at rest) and severity factor (0=no dystonia to 4=extreme/severe dystonia). Scores are weighted yielding a total score ranging from 0 to 120. The disability scale is a functional marker consisting of parental- or self-reported daily activities (involving speech, handwriting, feeding, eating, swallowing, hygiene, dressing, and walking), with scores ranging from 0 (completely independent) to 30 (completely dependent). A higher score indicates higher disease severity/disability.
Change from baseline to 6 months in disease-specific motor rating scale. For subjects with cervical dystonia, TWSTRS severity scale. | Baseline to 6 months
  The Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) severity subscale rates the severity of cervical dystonia. This scale consists of three subscales measuring symptom severity, disability, and pain. The severity scale is rated by the clinician and is composed of 11 items with a maximum score of 35. The disability and pain scales are patient-rated. The disability scale is composed of 6 items with a maximum score of 30. The pain scale is composed of 3 items with a maximum score of 20. The total TWSTRS score ranges from 0 to 85 points. Higher scores indicate higher severity/disability/pain.
Change from baseline to 1 year in disease-specific motor rating scale. For subjects with cervical dystonia, TWSTRS severity scale. | Baseline to 1 year
  The Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) severity subscale rates the severity of cervical dystonia. This scale consists of three subscales measuring symptom severity, disability, and pain. The severity scale is rated by the clinician and is composed of 11 items with a maximum score of 35. The disability and pain scales are patient-rated. The disability scale is composed of 6 items with a maximum score of 30. The pain scale is composed of 3 items with a maximum score of 20. The total TWSTRS score ranges from 0 to 85 points. Higher scores indicate higher severity/disability/pain.
Change from baseline to 2 years in disease-specific motor rating scale. For subjects with cervical dystonia, TWSTRS severity scale. | Baseline to 2 years
  The Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) severity subscale rates the severity of cervical dystonia. This scale consists of three subscales measuring symptom severity, disability, and pain. The severity scale is rated by the clinician and is composed of 11 items with a maximum score of 35. The disability and pain scales are patient-rated. The disability scale is composed of 6 items with a maximum score of 30. The pain scale is composed of 3 items with a maximum score of 20. The total TWSTRS score ranges from 0 to 85 points. Higher scores indicate higher severity/disability/pain.
Change from baseline to 3 years in disease-specific motor rating scale. For subjects with cervical dystonia, TWSTRS severity scale. | Baseline to 3 years
  The Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) severity subscale rates the severity of cervical dystonia. This scale consists of three subscales measuring symptom severity, disability, and pain. The severity scale is rated by the clinician and is composed of 11 items with a maximum score of 35. The disability and pain scales are patient-rated. The disability scale is composed of 6 items with a maximum score of 30. The pain scale is composed of 3 items with a maximum score of 20. The total TWSTRS score ranges from 0 to 85 points. Higher scores indicate higher severity/disability/pain.
Change from baseline to 4 years in disease-specific motor rating scale. For subjects with cervical dystonia, TWSTRS severity scale. | Baseline to 4 years
  The Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) severity subscale rates the severity of cervical dystonia. This scale consists of three subscales measuring symptom severity, disability, and pain. The severity scale is rated by the clinician and is composed of 11 items with a maximum score of 35. The disability and pain scales are patient-rated. The disability scale is composed of 6 items with a maximum score of 30. The pain scale is composed of 3 items with a maximum score of 20. The total TWSTRS score ranges from 0 to 85 points. Higher scores indicate higher severity/disability/pain.
Change from baseline to 5 years in disease-specific motor rating scale. For subjects with cervical dystonia, TWSTRS severity scale. | Baseline to 5 years
  The Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) severity subscale rates the severity of cervical dystonia. This scale consists of three subscales measuring symptom severity, disability, and pain. The severity scale is rated by the clinician and is composed of 11 items with a maximum score of 35. The disability and pain scales are patient-rated. The disability scale is composed of 6 items with a maximum score of 30. The pain scale is composed of 3 items with a maximum score of 20. The total TWSTRS score ranges from 0 to 85 points. Higher scores indicate higher severity/disability/pain.
Incidence of device- and procedure-related serious adverse events at 6 months | At 6 months
  Serious Adverse Events related to the device and procedure will be assessed.
  If the AE meets any of the criteria below, it is regarded as a serious adverse event (SAE).
  a) Led to a death, b) Led to a serious deterioration in health of the subject, that either resulted in i) a life-threatening illness or injury, or ii) a permanent impairment of a body structure or a body function, or iii) in-patient hospitalization or prolongation of existing hospitalization, or iv) medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function.
  v) chronic disease c) Led to fetal distress, fetal death or a congenital abnormality or birth defect.
Incidence of device- and procedure-related serious adverse events at 1 year | At 1 year
  Serious Adverse Events related to the device and procedure will be assessed.
  If the AE meets any of the criteria below, it is regarded as a serious adverse event (SAE).
  a) Led to a death, b) Led to a serious deterioration in health of the subject, that either resulted in i) a life-threatening illness or injury, or ii) a permanent impairment of a body structure or a body function, or iii) in-patient hospitalization or prolongation of existing hospitalization, or iv) medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function.
  v) chronic disease c) Led to fetal distress, fetal death or a congenital abnormality or birth defect.
Incidence of device- and procedure-related serious adverse events at 2 years | At 2 years
  Serious Adverse Events related to the device and procedure will be assessed.
  If the AE meets any of the criteria below, it is regarded as a serious adverse event (SAE).
  a) Led to a death, b) Led to a serious deterioration in health of the subject, that either resulted in i) a life-threatening illness or injury, or ii) a permanent impairment of a body structure or a body function, or iii) in-patient hospitalization or prolongation of existing hospitalization, or iv) medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function.
  v) chronic disease c) Led to fetal distress, fetal death or a congenital abnormality or birth defect.
Incidence of device- and procedure-related serious adverse events at 3 years | At 3 years
  Serious Adverse Events related to the device and procedure will be assessed.
  If the AE meets any of the criteria below, it is regarded as a serious adverse event (SAE).
  a) Led to a death, b) Led to a serious deterioration in health of the subject, that either resulted in i) a life-threatening illness or injury, or ii) a permanent impairment of a body structure or a body function, or iii) in-patient hospitalization or prolongation of existing hospitalization, or iv) medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function.
  v) chronic disease c) Led to fetal distress, fetal death or a congenital abnormality or birth defect.
Incidence of device- and procedure-related serious adverse events at 4 years | At 4 years
  Serious Adverse Events related to the device and procedure will be assessed.
  If the AE meets any of the criteria below, it is regarded as a serious adverse event (SAE).
  a) Led to a death, b) Led to a serious deterioration in health of the subject, that either resulted in i) a life-threatening illness or injury, or ii) a permanent impairment of a body structure or a body function, or iii) in-patient hospitalization or prolongation of existing hospitalization, or iv) medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function.
  v) chronic disease c) Led to fetal distress, fetal death or a congenital abnormality or birth defect.
Incidence of device- and procedure-related serious adverse events at 5 years | At 5 years
  Serious Adverse Events related to the device and procedure will be assessed.
  If the AE meets any of the criteria below, it is regarded as a serious adverse event (SAE).
  a) Led to a death, b) Led to a serious deterioration in health of the subject, that either resulted in i) a life-threatening illness or injury, or ii) a permanent impairment of a body structure or a body function, or iii) in-patient hospitalization or prolongation of existing hospitalization, or iv) medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function.
  v) chronic disease c) Led to fetal distress, fetal death or a congenital abnormality or birth defect.

CONTACTS AND LOCATIONS:
Overall Officials: Devyani Nanduri, Study Director — Abbott Medical Devices Neuromodulation
Locations (48):
- United States (23):
  - University of Aizona Health Sciences, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California at Davis, Sacramento, California
  - Colorado Neurodiagnostics, Littleton, Colorado
  - Neurosurgery One, Littleton, Colorado
  - University of Miami Hospital, Miami, Florida
  - University of South Florida - Department of Neurology, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Willis-Knighton Medical Center, Shreveport, Louisiana
  - Beth Israe Deaconess Medical Center, Boston, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical Center, Albany, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State Medical, Columbus, Ohio
  - Wright State University & Premier Health, Fairborn, Ohio
  - Center for Interventional Pain & Spine, Exton, Pennsylvania
  - Thomas Jefferson Department or Neurosurgery, Philadelphia, Pennsylvania
  - Allegheny General Hospital Department of Neurosurgery, Pittsburgh, Pennsylvania
  - Texas Movement Disorder Specialist, Georgetown, Texas
  - University of Utah Hospital, Salt Lake City, Utah
- Australia (2):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Melbourne Hospital - City Campus, Parkville, Victoria
- Helsinki University Central Hospital, Helsinki, Uusimaa, Finland
- France (4):
  - CHU Gabriel Montpied, Clermont-Ferrand, Auvergne
  - CHU de St Etienne, Saint-Etienne, Auvergne
  - Fondation Rothchild, Paris, ILE
  - CHU Hopital Pasteur, Nice, Provence-Alpes-Azur
- Germany (6):
  - Universitäts Klinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Medizinische Einrichtungen der Universität Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - UNIVERSITATSMEDIZIN der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
  - UKE Hamburg (Universitatsklinik Eppendorf), Hamburg
- Italy (3):
  - Az.Osp. Universitaria di Ferrara, Cona, Emilia-Romagna
  - Policlinico Universitario A. Gemelli, Rome, Lazio
  - Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta, Milan, Lombardy
- Spain (3):
  - Hospital Virgen de Rocio, Seville, Andalusia
  - Hospital Universitari Germans Trias I Pujol, Badalona, Catalonia
  - Hospital Universitario de la Princesa, Madrid
- Taiwan (2):
  - Chang Gung Memorial Hospital, Linkou District, Ntaiwan
  - Hualien Tzu Chi Hospital, Hualien City
- United Kingdom (4):
  - The Walton Centre, Liverpool, North West England
  - Southmead Hospita, Bristol, South West England
  - Queen Elizabeth University Hospital, Glasgow, Wdbtshr
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gharabaghi A, Groppa S, Casas E, Schnitzler A, Munoz-Delgado L, Marshall VL, Karl J, Zhang L, Alvarez R, Feldman MS, Soileau MJ, Luo L, Walter BL, Wu C, Lei H, Herz DM, Nanduri D, Salazar CA, Luca C, Weiss D. Real-world multicenter assessment of sustained clinical outcomes after digital deep brain stimulation. NPJ Digit Med. 2026 Jan 14. doi: 10.1038/s41746-025-02315-5. Online ahead of print. PMID 41535352